CLINICAL TRIAL: NCT01101594
Title: A Phase I/II Study of hLL1-DOX (Milatuzumab-Doxorubicin Antibody-Drug Conjugate) in Patients With Multiple Myeloma
Brief Title: A Study of hLL1-DOX (Milatuzumab-Doxorubicin Antibody-Drug Conjugate) in Patients With Multiple Myeloma
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Study was terminated due to lack of efficacy
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IM-T-hLL1-DOX-01
Record Dates: First submitted 2010-03-11; First posted 2010-04-12 (Estimated); Last update posted 2021-08-16 (Actual); Status verified 2020-03

CONDITIONS: Multiple Myeloma
Keywords: Treatment; Multiple Myeloma; Relapsed, refractory multiple myeloma
MeSH Terms: conditions — Multiple Myeloma; Recurrence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- hLL1-DOX (Experimental): 4 Different dose levels of hLL1-DOX will be studied in groups of 3-6 patients. Once an optimal dose has been found, up to additional 30 patients will be studied at that dose level.
  Interventions: Drug: hLL1-DOX (the doxorubicin conjugate of milatuzumab)

INTERVENTIONS:
Drug: hLL1-DOX (the doxorubicin conjugate of milatuzumab) — hLL1-DOX will be administered intravenously (through a vein) on days 1, 4, 8 & 11 every 21 days for up to 8 treatment cycles. 4 different dose levels of hLL1-DOX will be studied for safety and tolerability.
  Other Names: hLL1-DOX; Milatuzumab-DOX; CD74-DOX

SUMMARY:
This study is a Ph I trial to test the safety of the study drug, hLL1-DOX at different dose levels in patients with recurrent multiple myeloma. HLL1 is also known as milatuzumab and is attached to doxorubicin in this clinical trial.

DETAILED DESCRIPTION:
In this clinical research trial, hLL1-DOX will be administered on days 1, 4, 8 and 11. This treatment cycle will be repeated every 3 weeks as long as patients continue to tolerate it, for a maximum of 8 treatment cycles (approximately 6 months).

ELIGIBILITY:
Inclusion Criteria:

* Able to provide signed, informed consent;
* Male or female, >/= 18 years old;
* Multiple myeloma with one or more criteria for measurable disease (serum M protein > 0.5 gm/dl, urinary M protein excretion > 200 mg/24 hours, serum free light chain measurement >20 mg/dl,);
* Refractory or relapsed to at least two prior standard systemic anti-myeloma treatment regimens one of which must include either thalidomide, lenalidomide or bortezomib;
* Adequate performance status (Karnofsky Scale >/= 70%);
* Life expectancy at least 6 months;
* Adequate cardiac function: MUGA scan or 2D-ECHO with LVEF 55%, EKG with no medically relevant arrhythmia uncontrolled on medications;
* Adequate hematologic status within 2 weeks before study drug administration:
* Hemoglobin >/=8.0 g/dL and platelets >/=75,000/mm3 (both without transfusion or other hematologic support within 7 days of laboratory testing)
* White blood count (WBC) >/= 2,000/mm3and absolute neutrophil count (ANC) >/=1,500/mm3 (both without the use of colony stimulating factors within 7 days of laboratory testing);
* Adequate renal function: serum creatinine </+ 2.5 mg/mL;
* Adequate hepatic function
* AST and ALT </= 2.5 x the ULN
* Total bilirubin </= 1.5 x the ULN

Exclusion Criteria:

* 1. Pregnant or lactating women. Women of childbearing potential must have a negative pregnancy test Pregnancy testing is not required for post-menopausal or surgically sterilized women;
* Patients who are eligible for stem cell transplant.
* Women of childbearing potential and fertile men who are not practicing or who are unwilling to practice birth control while enrolled in the study until at least 12 weeks after the last hLL1-dox infusion;
* Prior local radiotherapy within 14 days; chemotherapy or kyphoplasty within 21 days, immunotherapy, plasmapheresis, or major surgery within 28 days; prior stem cell transplant within 12 weeks.
* Must have no persistent ≥ Grade 2 toxicity from prior treatments;
* Prior treatment with any other therapeutic agents for MM or investigational agents within 4 weeks, unless off study, and agreed by Sponsor;
* A history of allergic or adverse reactions to anthracycline/anthracenedione agents;
* Cumulative life-time anthracycline/anthracenedione exposure exceeding 300 mg/m2 (including daunorubicin, idarubicin, epirubicin or mitoxantrone);
* Known to be HIV positive, or any prior hepatitis B or C infection;
* Any history of clinically significant autoimmune disease (e.g., collagen vascular disorders, autoimmune hepatitis, Coombs positive anemia/thrombocytopenia, etc.)
* Prior history of mediastinal or pericardial external beam radiation therapy.
* Prior history of treatment with trastuzumab, unless discussed with and agreed to by Medical Monitor.
* Systemic infection or requiring anti-infectives within 7 days before first dose of study drug;
* Substance abuse or other concurrent medical conditions that, in the Investigator's opinion, could confound study interpretation or affect the patient's ability to tolerate or complete the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2010-07; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
All patients administered any dose of study drug will be included in the evaluation of safety | Before infusion, 5 min after start, every 15 min until completion, then 30, 60, 90 and 120 min later of each dose of study drug
  The frequency and severity of adverse events (AEs) will be tabulated by MedDRA Preferred Term and System Organ Class (SOC) for each dose group. AEs will be classified using the MedDRA version 8.0 with severity assessed by NCI CTC v3 toxicity grades

SECONDARY OUTCOMES:
Determine the therapeutic efficacy of hLL1-DOX in this patient population | During treatment and the changes at 4, 8 and 12 weeks after treatment and then every 3 months for up to 2 years
  All patients who were treated with at least one complete dose of study drug and have available response assessment data will constitute the efficacy population. For efficacy evaluations, treatment responses based on IMWG Response Criteria, response duration and progression-free survival will be tabulated and summarized by descriptive statistics for patients in each dose group.

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - MD Anderson Orlando, Orlando, Florida
  - Georgia Cancer Specialists, Atlanta, Georgia
  - Hackensack University Medical Center, Hackensack, New Jersey
  - University Hospital of Pennsylvania, Philadelphia, Pennsylvania
  - MD Anderson Center, Houston, Texas

REFERENCES:
- [Background] Griffiths GL, Mattes MJ, Stein R, Govindan SV, Horak ID, Hansen HJ, Goldenberg DM. Cure of SCID mice bearing human B-lymphoma xenografts by an anti-CD74 antibody-anthracycline drug conjugate. Clin Cancer Res. 2003 Dec 15;9(17):6567-71. PMID 14695162
- [Background] Burton JD, Ely S, Reddy PK, Stein R, Gold DV, Cardillo TM, Goldenberg DM. CD74 is expressed by multiple myeloma and is a promising target for therapy. Clin Cancer Res. 2004 Oct 1;10(19):6606-11. doi: 10.1158/1078-0432.CCR-04-0182. PMID 15475450
- [Background] Pawlak-Byczkowska EJ, Hansen HJ, Dion AS, Goldenberg DM. Two new monoclonal antibodies, EPB-1 and EPB-2, reactive with human lymphoma. Cancer Res. 1989 Aug 15;49(16):4568-77. PMID 2663143
- [Background] Stein R, Gupta P, Chen X, Cardillo TM, Furman RR, Chen S, Chang CH, Goldenberg DM. Therapy of B-cell malignancies by anti-HLA-DR humanized monoclonal antibody, IMMU-114, is mediated through hyperactivation of ERK and JNK MAP kinase signaling pathways. Blood. 2010 Jun 24;115(25):5180-90. doi: 10.1182/blood-2009-06-228288. Epub 2010 Jan 25. PMID 20101022
- [Background] Sapra P, Stein R, Pickett J, Qu Z, Govindan SV, Cardillo TM, Hansen HJ, Horak ID, Griffiths GL, Goldenberg DM. Anti-CD74 antibody-doxorubicin conjugate, IMMU-110, in a human multiple myeloma xenograft and in monkeys. Clin Cancer Res. 2005 Jul 15;11(14):5257-64. doi: 10.1158/1078-0432.CCR-05-0204. PMID 16033844
- [Background] Stein R, Mattes MJ, Cardillo TM, Hansen HJ, Chang CH, Burton J, Govindan S, Goldenberg DM. CD74: a new candidate target for the immunotherapy of B-cell neoplasms. Clin Cancer Res. 2007 Sep 15;13(18 Pt 2):5556s-5563s. doi: 10.1158/1078-0432.CCR-07-1167. PMID 17875789
- [Background] Mark T, Martin P, Leonard JP, Niesvizky R. Milatuzumab: a promising new agent for the treatment of lymphoid malignancies. Expert Opin Investig Drugs. 2009 Jan;18(1):99-104. doi: 10.1517/13543780802636162. PMID 19053886
- [Background] Stein R, Smith MR, Chen S, Zalath M, Goldenberg DM. Combining milatuzumab with bortezomib, doxorubicin, or dexamethasone improves responses in multiple myeloma cell lines. Clin Cancer Res. 2009 Apr 15;15(8):2808-17. doi: 10.1158/1078-0432.CCR-08-1953. Epub 2009 Apr 7. PMID 19351768